CLINICAL TRIAL: NCT00090909
Title: A Phase II Study Of Gemcitabine, Cisplatin, and Dexamethasone In Patients With Relapsed Or Refractory Hodgkin Lymphoma
Brief Title: Gemcitabine, Cisplatin, and Dexamethasone in Treating Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000380845; UCLA-030402301; LILLY-B9E-US-X394
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Cisplatin; Dexamethasone; Gemcitabine

INTERVENTIONS:
Drug: cisplatin
Drug: dexamethasone
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, cisplatin, and dexamethasone, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine and cisplatin together with dexamethasone works in treating patients with relapsed or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and maximum response in patients with relapsed or refractory Hodgkin's lymphoma treated with gemcitabine, cisplatin, and dexamethasone.
* Determine time to progression in patients treated with this regimen who are not undergoing stem cell transplantation.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is an open-label study.

Patients receive gemcitabine IV over 1 hour on days 1 and 8, cisplatin IV over 3 hours on day 1, and oral dexamethasone twice daily on days 1-4. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed until disease progression.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Hodgkin's lymphoma
* Measurable disease by radiological or clinical findings
* Failed at least 1, but no more than 2, prior standard chemotherapy regimens

  * High-dose chemotherapy administered after a chemotherapy course is considered 2 courses
* No evidence of CNS disease
* No history of myelodysplastic syndromes

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC > 2,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 75,000/mm^3
* Hemoglobin > 8.0 g/dL

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* AST and ALT < 5 times ULN

Renal

* Creatinine < 1.5 times ULN

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior gemcitabine
* More than 6 months since prior high-dose chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2003-06; Primary Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States